CLINICAL TRIAL: NCT00808197
Title: Choroidal Blood Flow and Progression of Age-Related Macular Degeneration in the Fellow Eye in Patients With Unilateral Choroidal Neovascularisation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OPHT-140501
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Last update posted 2008-12-15 (Estimated); Status verified 2008-12

CONDITIONS: Regional Blood Flow
Keywords: AMD; choroidal blood flow; fellow eye in patients with unilateral choroidal neovascularisation

ARMS (1):
- 1 (Experimental): Observatory, longitudinal, 3-years follow up study
  Interventions: Procedure: ocular blood flow measurement

INTERVENTIONS:
Procedure: ocular blood flow measurement — Ocular blood flow will be determined by non-invasive methods, including laser Doppler flowmetry and laser interferometry

SUMMARY:
Age-related macular degeneration (AMD) is the chief cause of severe and irreversible loss of vision in developed countries. The prevalence of AMD increases dramatically with age.

The early stage (or dry AMD) is associated with minimal visual impairment and is characterized by large drusen and pigmentary abnormalities in the macula. The late stage is a neovascular, exudative form. This so called exudative AMD includes serous or hemorrhagic detachment of retinal pigment epithelium and choroidal neovascularization leading to severe loss of vision (20/200 or worse). Patients with unilateral CNV (choroidal neovascularisation) have a significant risk of CNV developing in the second eye.

Choroidal blood flow is of great importance for normal visual function. Several reports have provided evidence suggesting that choroidal blood flow is decreased in subjects with AMD. In late stages of AMD angiogenesis leads to the formation of choroidal neovascularization that can cause severe visual impairment by disrupting normal macular function.

The purpose of this evaluation is to investigate a possible link between alterations in choroidal blood flow and the development of CNV and serous detachment in the fellow eye of patients with AMD and unilateral neovascular maculopathy. This longitudinal study may provide important findings with respect to natural history and visual prognosis of patients with neovascularized AMD.

Ocular blood flow will be determined by non-invasive methods, including laser Doppler flowmetry and laser interferometry

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with unilateral choroidal neovascular AMD and 2-4 risk factors for AMD in the fellow eye.
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant Ametropy < 4 dpt.

Exclusion Criteria:

* Abuse of alcoholic beverages
* Participation in a clinical trial in the 3 weeks preceding the study
* Any signs of diabetic retinopathy
* Glaucoma
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Estimated)

PRIMARY OUTCOMES:
Choroidal blood flow (laser Doppler flowmetry)
Fundus pulsation amplitude (laser interferometry)

CONTACTS AND LOCATIONS:
Overall Officials: Leopold Schmetterer, Prof. Dr., Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria